CLINICAL TRIAL: NCT02860728
Title: A Novel Individualized Resistance Training Program to Prehabilitate Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Resistance Training to Prehabilitate Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Eves, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H16-01019
Record Dates: First submitted 2016-08-05; First posted 2016-08-09 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Resistance Training; Exercise Training; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

ARMS (1):
- Resistance training (Experimental): Patients with COPD will participate in 4 weeks (12 sessions) of individualized, non-linear, lower body resistance training.
  Interventions: Behavioral: Individualized Resistance Training

INTERVENTIONS:
Behavioral: Individualized Resistance Training — Lower body resistance exercises will be prescribed in various combinations over multiple days and individually modified and progressed to achieve advances in both movement pattern, intensity, and exercise volume.

SUMMARY:
Structural changes in skeletal muscles of patients with chronic obstructive pulmonary disease (COPD) have been linked to impaired muscle function, reduced exercise capacity, and increased mortality associated with this disease. Muscle dysfunction also contributes to dyspnea intensity and the ability to sustain exercise, making aerobic exercise training intolerable at the intensity and/or volume required to achieve clinically important changes. Resistance training (RT) is an attractive exercise modality because it is efficacious and more tolerable initially. No work has examined whether a short-term RT program can reduce exertional symptoms and improve exercise tolerance (dyspnea and leg fatigue) in patients with COPD.

DETAILED DESCRIPTION:
Skeletal muscle dysfunction is common in patients with COPD and has been recognized as a contributing factor to reduced exercise capacity, health related quality of life and increased mortality associated with this disease. Several structural changes in the limb muscles of patients have previously been reported and have been linked to the known reductions in muscle strength and endurance commonly reported in COPD. Muscle dysfunction, lower extremity muscle strength, and muscle fatigue also contribute to the intensity of dyspnea and the ability to sustain exercise mostly through stimulation of type III and IV muscle afferents. As such, many patients who primarily perform aerobic exercise training as part of pulmonary rehabilitation are unable to tolerate the intensity and/or volume of exercise required to achieve clinically important changes in exercise capacity or symptom relief. Resistance training (RT) is an attractive exercise modality for patients with COPD because it is efficacious and often more tolerable initially. To our knowledge no one has examined whether similar benefits to those elicited by longer RT programs can be attained in just 4 weeks using multi-joint, multi-muscle exercises and individualized progression. If a short term RT program can improve muscle quality, enhance endurance, and reduce type III and IV afferent activity then it would reduce the drive to breathe and thus dyspnea. These adaptations would likely translate into improved exercise tolerance making it feasible to "pre-habilitate" COPD patients with tolerable RT, allowing them to achieve a higher volume/intensity of endurance training, thus making pulmonary rehabilitation more effective.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers >6 months
* FEV1/FVC <0.7 and lower limit of normal
* 30%< FEV1 pred <70%
* Stable (no exacerbation for >3 months)

Exclusion Criteria:

* Cardiovascular and cerebrovascular disease
* Diabetes
* Cardiovascular contraindications to exercise
* Uncontrolled hypertension
* Currently performing regular structured exercise >3x/week for 30 minutes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Dyspnea | Baseline and post 4 weeks (12 sessions) of resistance training
  The change in the sensory intensity of dyspnea measured at an iso-time during the constant load exercise trials post RT

SECONDARY OUTCOMES:
Exercise Tolerance | Baseline and post 4 weeks (12 sessions) of resistance training
  The change in the time to exhaustion during constant load exercise on a stationary cycle ergometer.
Secondary Dyspnea Outcomes | Baseline and post 4 weeks (12 sessions) of resistance training
  The change in the unpleasantness and sensory qualities of dyspnea measured at an iso-time during the constant load exercise trials post RT
Quadriceps Fatigue | Baseline and post 4 weeks (12 sessions) of resistance training
  Change in the amount of decline in force production after 3 minutes of electrical stimulation of femoral nerve at 25% of maximal voluntary contraction
Muscle Strength and Endurance | Baseline and post 4 weeks (12 sessions) of resistance training
  The change in 6RM quadriceps muscle strength and quadricep muscle endurance at 50% of predicted 1 RM

CONTACTS AND LOCATIONS:
Overall Officials: Neil Eves, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada